CLINICAL TRIAL: NCT04619355
Title: Korean Near-infrared Spectroscopy(NIRS)-Intravascular Ultrasound (IVUS) Multicenter Registry: a Comprehensive Study
Brief Title: Korean NIRS-IVUS Multicenter Registry
Status: Recruiting | Type: Observational
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Soon Jun Hong, Professor, Korea University Anam Hospital
Other Study IDs: NIRS-IVUS in Korea
Record Dates: First submitted 2020-11-02; First posted 2020-11-06 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Coronary Artery Disease With Myocardial Infarction
Keywords: NIRS; IVUS
MeSH Terms: conditions — Coronary Artery Disease, Autosomal Dominant, 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- TVC K-Registry
  Interventions: Device: NIRS-IVUS

INTERVENTIONS:
Device: NIRS-IVUS — Near-infrared spectroscopy-intravascular ultrasound can be implemented in parallel with intravascular ultrasound and provides important information for predicting prognosis by measuring the lipid component of atherosclerotic plaques.

SUMMARY:
Heart diseases known as the second cause of death in Koreans are coronary artery diseases such as angina and myocardial infarction. Coronary artery disease occurs when fat components, such as cholesterol, accumulate in the body. When these fat components are deposited in blood vessels, blood vessels' walls become thick, and the blood vessels narrow, which interferes with circulation. Without smooth circulation, the heart muscle does not function properly because the supply of oxygen and nutrient-rich blood, which is necessary for the heart to function normally, is not properly supplied. It leads to angina pectoris and chest pain and can cause myocardial infarction or even heart attack. Coronary artery disease in various aspects has a high mortality rate when it occurs in old age. The methods currently used for diagnosis and treatment are coronary angiography, percutaneous coronary intervention (PCI), and myocardial partial blood flow reserve history. There is a wide variety of tests (Fractional Flow Reserve, FFR), near-infrared spectroscopy intravascular ultrasound (NIRS-IVUS).

In addition to the various aspects and treatment methods of this disease, treatment is often difficult, so the clinical significance is great. In the case of PCI, one of the methods of examination and treatment, the National Cardiovascular Data Registry (NCDR) has been established to establish guidelines for improving patient prognosis after surgery in the United States. NCDR, which started with the American College of Cardiology (ACC) initiative, is currently in an indispensable position for establishing clinical practice guidelines such as monitoring treatment-related indicators, quality improvement (QI), and clinical research. In charge. Besides, in recent years, the use of new drugs or new devices (Post-Market Surveillance), real-time risk estimation, and personalized planning is increasing.

Research to analyze the prognosis of various aspects of coronary artery disease, tests, and procedures has been constantly conducted, but comprehensive studies that can be used to improve the overall treatment are considered to be insufficient. At this point, a comprehensive study is required to establish clinical guidelines and to develop them continuously.

In particular, the area that needs research is whether or not future events can be prevented using vascular imaging. Studies have shown that if lipids are actively treated with statins, the lipid component of atherosclerotic plaques can be significantly reduced in just a few weeks. Suggests. According to the results of a YELLOW (Reduction in Yellow Plaque by Aggressive Lipid-Lowering Therapy) study published in 2012 based on a near-infrared spectroscopy-vascular ultrasound analysis, the active treatment group of statins showed the lipid-core burden index compared to the standard treatment group. ) showed a significant decrease.

Accordingly, this study collects all comprehensive indicators such as test methods, test results, procedures, and treatment results for all patients undergoing near-infrared spectroscopy-vascular ultrasound treatment in Korea, including this institution, A comprehensive study of the disease registry related to the near-infrared spectroscopy-vascular ultrasound procedure is conducted to determine the type of disease, the number of affected vessels, and disease-related indicators.

ELIGIBILITY:
Inclusion Criteria:

* patient who underwent PCI using NIRS-IVUS
* Subjects who agreed to the study plan and clinical follow-up plan, voluntarily decided to participate in this clinical study and agreed in writing to the subject consent form

Exclusion Criteria:

* Subjects who cannot perform cardiovascular angiography due to severe symptoms of heart failure
* Subjects whose expected life expectancy is within 1 year due to the accompanying disease
* Women of childbearing age who plan to become pregnant within the study period

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Since this study includes all inpatients who have undergone near-infrared spectroscopy-intravascular ultrasonography, the target number of subjects is not limited, and all patients suitable for the study will be enrolled. After the end of the study, the total number of institutional procedures will be finalized to calculate the number of enrolled subjects.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2010-01-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Cardiac death | 1 Day
  Cardiac death

SECONDARY OUTCOMES:
MACE | 1 Day
  Composite of cardiac death, MI, unstable angina or progressive angina either requiring revascularization or with rapid lesion progression
Death | 1 Day
  Any cause of death
Stent thrombosis | 1 Day
  Stent thrombosis
Stroke | 1 Day
  Stroke

CONTACTS AND LOCATIONS:
Overall Officials: Soon Jun Hong, MD, PhD, Principal Investigator — Korea University Anam Hospital
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea